CLINICAL TRIAL: NCT02690857
Title: Efficacy of Docosahexanoic Acid on Lipid Peroxidation in Subjects With Cystic Fibrosis
Brief Title: Study of Docosahexanoic Acid in Patients With Cystic Fibrosis (CF)
Acronym: OMEGAMUCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008.533
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2016-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Docosahexaenoic Acids; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Docosahexaenoic acid (Experimental): Each capsule of DHA contains 100 mg DHA in triglycerides from algal oil, 0.125 mg alpha-tocopherol and 0.125 mg ascorbic acid.
  Subjects receive an orally and daily ingestion of DHA capsules (5mg/kg for 15 days followed by 10 mg/kg for another 15 days without interruption between the 2 periods).
  Interventions: Drug: Docosahexaenoic acid
- Sunflower oil (Placebo Comparator): Placebo capsules contain the same quantities of antioxidants and triglycerides of sunflower oil. Subjects receive an orally and daily ingestion of placebo capsules for 28 days.
  Interventions: Drug: Sunflower Oil

INTERVENTIONS:
Drug: Docosahexaenoic acid
  Arms: Docosahexaenoic acid
Drug: Sunflower Oil
  Arms: Sunflower oil

SUMMARY:
Patients with Cystic Fibrosis have increased oxidative stress and impaired antioxidant systems. Under certain conditions, docosahexaenoic acid (DHA) intake may have a favorable role in reducing redox status.

In this randomized, double-blind, cross-over study, DHA (Pro-Mind) and placebo (sunflower oil) capsules, will be given, daily to 10 patients, 5 mg/kg for 2 weeks then 10 mg/kg for the next 2 weeks. Biomarkers of lipid peroxidation and vitamin E levels will be measured. Plasma and platelet lipid compositions will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male with confirmed diagnosis of Cystic Fibrosis with a sweat chloride > 60 mmol/L and a pancreatic insufficiency.
* Subjects will be aged between 6 and 18 years and be prepubescent, or aged between 18 and 30 years
* Body weight > 26 kg
* Stable CF disease as judged by the investigator.
* Subjects must have an Forced Expiratory Volume at one second > 40 % of predicted normal for age, sex and height at the screening visit.
* Subjects should not have enteral or parenteral nutrition.
* No periodic IV lipidic emulsion administration. Subjects must not consume food supplements rich in OMEGA-3 on a regular basis.

Exclusion Criteria:

* Subjects with cirrhosis and portal hypertension.
* Subjects with Cystic fibrosis related diabetes.
* Concomitant participation in another clinical study.
* Known allergy or intolerance to the active principle.
* Subjects with major blood coagulation anomalies, patients under anticoagulants or aspirin (long term therapy).
* Subjects on a transplant waiting list.

Ages: 6 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in 8-isoprostane level in urine. | Day 14
  Measured by urinalysis (Immunoassay).

SECONDARY OUTCOMES:
Change in 11-dehydro-thromboxane B2 in urine. | Day 28
  Measured by urinalysis (Immunoassay).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 28
  Measured by vital signs
Change in percent predicted forced expiratory volume in 1 second | from baseline through Day 28
  Spirometry
Evaluation of the effect of DHA on specific biomarkers. | Day 28
  Gas chromatography, immunoassays, fluorimetry. (in plasma : lipids, vitamin E and in platelet : lipids, vitamin E, thromboxane B2, malondialdehyde).

REFERENCES:
- [Result] Vericel E, Mazur S, Colas R, Delaup V, Calzada C, Reix P, Durieu I, Lagarde M, Bellon G. Moderate intake of docosahexaenoic acid raises plasma and platelet vitamin E levels in cystic fibrosis patients. Prostaglandins Leukot Essent Fatty Acids. 2016 Dec;115:41-47. doi: 10.1016/j.plefa.2016.10.008. Epub 2016 Oct 18. PMID 27914512